CLINICAL TRIAL: NCT02901379
Title: Effect of 80-mg Atorvastatin on Myocardial Edema Following Coronary Artery Bypass Surgery in Relation With Follistatin-Like Protein-1
Brief Title: Effect of 80-mg Atorvastatin on Myocardial Edema
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cardiovascular Center Harapan Kita Hospital Indonesia (Other)
Responsible Party: Principal Investigator, Rita Zahara, Cardiologist, National Cardiovascular Center Harapan Kita Hospital Indonesia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LB.02.01/VII/090/KEP.013/2016
Record Dates: First submitted 2016-09-06; First posted 2016-09-15 (Estimated); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Myocardial Edema
Keywords: atorvastatin; myocardial edema; Follistatin-like 1; FSTL1; atorvastatin 80mg; coronary artery bypass surgery
MeSH Terms: interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atorvastatin 80mg (Experimental): Subjects who will receive atorvastatin 80mg for two weeks
  Interventions: Drug: Atorvastatin 80mg
- Atorvastatin 10mg (Active Comparator): Subject who will receive atorvastatin 10mg
  Interventions: Drug: Atorvastatin 10mg

INTERVENTIONS:
Drug: Atorvastatin 80mg — Subject will be given atorvastatin 80mg for two weeks
  Other Names: Lipitor
  Arms: Atorvastatin 80mg
Drug: Atorvastatin 10mg — Subjects will be give atorvastatin 10mg as part of standard therapy in hospital
  Other Names: Lipitor
  Arms: Atorvastatin 10mg

SUMMARY:
The purpose of this study is to determine whether atorvastatin 80mg can reduce the development of myocardial edema following coronary artery bypass surgery.

This study also want to determine:

1. whether atorvastatin 80mg can influence Follistatin-like 1 (FSTL1) plasma level following bypass surgery?
2. whether there is correlation between myocardial edema and FSTL1 plasma level?
3. the efficacy of atorvastatin 80mg compared to atorvastatin 10mg in reducing hs-CRP (high sensitive-C reactive protein) and MDA (malondialdehyde) plasma level following bypass surgery?
4. the efficacy of atorvastatin 80mg compared to atorvastatin 10mg in raising PKA and PKB plasma level following bypass surgery?

DETAILED DESCRIPTION:
This study is an double blinded experimental study using parallel design. Study subjects are patients in Harapan Kita hospital who are registered to CABG (Coronary Artery Bypass Graft) surgery and fulfill all the eligibility criteria.

The subjects will be first consecutively selected, with male age 40-65 as the criteria. After that the investigators do the randomization with block randomization method. All the subjects will be given drug with label A and label B (only the pharmacist know the which dose of atorvastatin belong to which label).

Total subjects needed for this study are 30 (15 belong to study group and 15 belong to control group) MRI (Magnetic Resonance Imaging) results will be read by two radiologists, and analyzed using cronbach alpha. The results are considered equal if the cronbach >0,7. If it is proven to be unequal, then the third radiologist will decide.

Statin is known to have several adverse effects, such as myopathy, myositis to rhabdomyolysis, elevated liver enzyme, memory loss, GI (gastrointestinal) disturbance, and severa others. Therefore, the investigators will check baseline CK (creatine kinase) and liver enzyme at the beginning of the study, before the surgery, and if the patient feel any symptoms. Statin will be stopped if patient decide to stop, or if there is increase in ALT (alanine aminotransferase) higher that three time upper normal value, or if there is increase in CK higher than ten times upper normal value.

Statistical analysis using IBM SPSS statistics version 21.0. Comparative analysis for variables such as smoking history, obesity, hypertension, dyslipidemia, diabetes, family history, infarct history, ACE-I/ARB (angiotensin converting enzyme inihibitor /angiotensin receptor blocker) therapy will be using chi-square or fischer. Comparative analysis for variables T2 relaxation time, FSTL1, hs-CRP, PKA (protein kinase A), PKB (Protein Kinase B), MDA, age, CPB (Cardiopulmonary Bypass) time, CABG time will using unpaired t-test or Mann-whitney. Correlative analysis between FSTL1 and T2 relaxation time will be using Pearson test.

ELIGIBILITY:
Inclusion Criteria:

* Patients with coronary artery disease indicated for CABG surgery
* has signed informed consent

Exclusion Criteria:

* high risk EURO (European System for Cardiac Operative Risk Evaluation) score
* creatinin value>2 g/dl
* direct bilirubin value >3 mg/ml
* AST/ALT (aspartate transaminase / alanine transaminase) value >1,5 times UNL (upper normal limit)
* high pre-operative CKMB (Creatine Kinase-MB) and troponin
* LVEF (Left Ventricular Ejection Fraction) <45%
* concomitant valve disease required surgery
* contraindicated for MRI
* high degree ventricular arrhytmia
* coagulation disorder
* COPD (chronic obsructive pulmonary disease)
* HIV (Human Immunodeficiency Virus) +, HBV (Hepatitis B Virus)+, HCV (Hepatitis C Virus) +
* conduction abnormality, pacemaker
* electrolyte or blood gas disturbance
* receiving immunosuppressive drug or cytotoxic agent 4 weeks before surgery
* receiving macrolide, azole antifungal, fibrate, or protease inhibitor HIV drug

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-10; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
T2 relaxation time | day 6 after CABG
  T2 relaxation time (in ms) difference between control and study group

SECONDARY OUTCOMES:
FSTL1 plasma level | day 6 after CABG
  FSTL1 plasma level difference between control and study group
PKA plasma level | day 6 after CABG
  PKA plasma level difference between control and study group
PKB plasma level | day 6 after CABG
  PKB plasma level difference between control and study group
hs-CRP plasma level | day 1 after CABG
  hs-CRP plasma level difference between control and study group
MDA plasma level | day 1 after CABG
  MDA plasma level difference between control and study group
Change from baseline FSTL1 plasma level | day 1 and day 6 after CABG
Change from baseline PKA plasma level | day 1 and day 6 after CABG
Change from baseline PKB plasma level | day 1 and day 6 after CABG

CONTACTS AND LOCATIONS:
Overall Officials: Rita Zahara, Principal Investigator — National Cardiovascular Center Harapan Kita

IPD SHARING:
Plan to Share IPD: No